CLINICAL TRIAL: NCT05475210
Title: Phase I, Open-Label Study of the Safety and Dosimetry of a 3-Dose Regimen of Escalating Doses of 177Lu-DOTA-EB-TATE in Adult Patients With Advanced, Well- Differentiated Neuroendocrine Tumors
Brief Title: 177Lu-DOTA-EB-TATE in Adult Patients With Advanced, Well- Differentiated Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Molecular Targeting Technologies, Inc. (Industry)
Collaborators: ClinSmart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTTI-EBT-001; 21-362 (Other: Memorial Sloan-Kettering Cancer Center IRB)
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — (177)Lu-DOTA-EB-TATE; amino-acid, glucose, and electrolyte solution

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Peptide Receptor Radionucleotide Therapy (PRRT) (Experimental): The treatment regimen will consist of a single-dose intravenous administration of 177Lu-DOTA-EB-TATE per 6-week cycle, for a total of 2 cycles. The dose per cycle will be fixed for each patient and will be escalated in 3 different dose levels, from 50 mCi to 150 mCi (1.85 -5.55 GBq). Each dose of 177Lu-DOTA-EB-TATE will be administered in association with intravenous renal protective amino acid solutions.
  Interventions: Drug: 177Lu-DOTA-EB-TATE; Other: Amino Acid Solution

INTERVENTIONS:
Drug: 177Lu-DOTA-EB-TATE — Peptide Receptor Radionucleotide Therapy ( PRRT) using 177Lu-DOTA-EB-TATE with a defined number of cycles will be administered.
Other: Amino Acid Solution — The Amino acid solution to be used in this study will contain a mixture of lysine and arginine diluted in an electrolyte solution.
  Other Names: Arginine-Lysine Solution

SUMMARY:
This is a Phase I clinical trial to assess the safety and dosimetry profiles of 177Lu-DOTA-EB-TATE in patients with advanced, metastatic or inoperable, somatostatin receptor-positive, well-differentiated GEP-NETs.

ELIGIBILITY:
Inclusion Criteria:

Ability to understand and willing to sign a written informed consent document

Aged 18 years or older

Histologically proven or cytologically confirmed, inoperable, GEP-NETs

Neuroendocrine tumors (NETs) of grade 1, 2 and 3 according to World Health Organization (WHO) 2017 classification

Measurable disease as defined by Response Criteria in Solid Tumors (RECIST) version 1.1

Overexpression of somatostatin receptors of the target lesions in 68Ga-DOTA-TATE positron emission tomography (PET)/computed tomography (CT) with SUV of lesions greater than normal liver in at least 1 lesion

A Cockcroft Gault calculated creatinine clearance > 60 mL/min

Karnofsky performance status scale ≥ 70%

Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation, including follow-up (7 months after the last dose of study drug for women and 4 months for men).

Previous local therapy (e.g., chemoembolization or bland embolization) is allowed if completed >4 weeks prior to study entry.

Previous surgery no less than 6 weeks prior to study entry.

Either no prior treatment with 177Lu-DOTA-TATE or at least 12 months progression-free survival (PFS) after prior treatment with 177Lu-DOTA-TATE

Exclusion Criteria:

Women who are pregnant or breastfeeding

History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-DOTA-EB-TATE as assessed from medical records

Previous treatment with more than 4 cycles of 177Lu-DOTA-TATE

Participant has had prior chemotherapy, targeted cancer therapy, immunotherapy, or treatment with an investigational anticancer agent within 4 weeks or 4 half-lives whichever is longer, before the first administration of study drug.

Participant has not fully recovered from major surgery or significant traumatic injury prior the first dose of study drug or expects to have major surgery during the study period or within 3 months after the last dose of study drug.

Life expectancy < 6 months as assessed by the treating physician

> 80% liver involvement by tumor

> 25% bone marrow involvement by tumor

Poorly differentiated neuroendocrine neoplasms, such as poorly differentiated neuroendocrine carcinoma, small- and large-cell neuroendocrine carcinoma; mixed neuroendocrine-non-neuroendocrine neoplasm (MiNEN); Grade 3 neuroendocrine carcinomas (NEC)

Presence of somatostatin receptor negative lesions if they cannot be addressed with loco-regional therapies prior to the treatment start

Deteriorated renal function, as indicated by a serum creatinine clearance > 1.7 mg/dL

Deteriorated bone marrow function

Deteriorated liver function

Toxicities from prior therapies that have not resolved to grade 1 or grade 0

Active and clinically significant bacterial, fungal, or viral infection, including hepatitis B (HBV), hepatitis C (HBC), know human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness

Known brain metastases and/or carcinomatous meningitis, unless these metastases have been treated and stabilized

Uncontrolled diabetes mellitus as defined by a HbA1c >9%

Impossibility to interrupt short-acting octreotide for 24 h before and 24 h after the administration of 177Lu-DOTA-EB-TATE; impossibility to have an interval of ≥4 weeks between octreotide and 177Lu-DOTA-EB-TATE

The use of somatostatin and its analogues within 4 months of a planned 177Lu-DOTA-EB-TATE treatment

Uncontrolled, intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Prior external beam radiation therapy involving >25% of the bone marrow

Unmanageable urinary incontinence rendering the administration of 177Lu-DOTA-EB-TATE unsafe

Other known co-existing malignancies except non-melanoma skin cancer and carcinoma in situ of the uterine cervix, unless definitively treated and with no evidence of recurrence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2022-06-18 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of 177Lu-DOTA-EB-TATE assessed from the number of patients with treatment-related adverse events. | 16-17 months
To identify the dose-limiting toxicities (DLTs) of escalating doses of 177Lu-DOTA-EB-TATE up to 150 mCi. | 16-17 months
To determine if the maximum tolerated dose is among the explored doses of 50, 100 and 150 mCi. | 16-17 months

SECONDARY OUTCOMES:
To evaluate the differential safety of 177Lu-DOTA-EB-TATE, expressed as the number of patients with treatment-related adverse events following 177Lu-DOTA-EB-TATE. | 16-17 months
To evaluate dosimetry levels in patients following 2 cycles of 177Lu-DOTA-EB-TATE. | 16-17 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bodei, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No